CLINICAL TRIAL: NCT05682560
Title: A Randomized Controlled Phase IIa, Two-arm Study to Assess the Safety and Efficacy of Human Umbilical Cord Blood (RegeneCyte) Infusion in Patients with Post-COVID Syndrome
Brief Title: Human Umbilical Cord Blood (RegeneCyte) Infusion in Patients with Post-COVID Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: StemCyte, Inc. (Industry)
Collaborators: StemCyte Taiwan Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: StemCyte International, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCUS001
Record Dates: First submitted 2023-01-11; First posted 2023-01-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Long COVID; Post-COVID Syndrome; Post COVID-19 Condition
Keywords: Long COVID; Post-COVID Syndrome; Post-COVID condition; Umbilical cord blood; RegeneCyte
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- REGENECYTE (Experimental): HPC, Cord Blood
  Interventions: Biological: REGENECYTE
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: REGENECYTE — HPC, Cord Blood
  Arms: REGENECYTE
Biological: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
REGENECYTE (HPC, Cord Blood, hUCB) for treatment in patients with post-COVID.

DETAILED DESCRIPTION:
This is a two-arm, single-center, single-blind, randomized, placebo-controlled phase IIa study. A total of 30 subjects with post-COVID will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged ≥ 18
* 2. With post-COVID syndrome
* 3. Has had a recent (within 7 days) negative SARS-CoV-2 test (an approved PCR or antigen test)
* 4. Able to provide signed informed consent (by the subject or his/her legally authorized representative)
* 5. Is willing and able to participate in all aspects of the study, including completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing a written informed consent

Exclusion Criteria:

* 1. Neurological disorders prior to COVID-19 diagnosis
* 2. With pre-existing terminal illness
* 3. With known immune disease
* 4. Is pregnant or breastfeeding
* 5. Is currently participating in another investigational study or has been taking any other investigational product within the last 4 weeks before screening
* 6. Has received any vaccination within 3 weeks prior to the first IP infusion
* 7. Judged by the investigator to be not suitable for study participation
* 8. Under the conditions that may increase risk of complications based on the medical judgment of the investigator and the parameters

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Baseline to Week 26
  Incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Change of fatigue score as measured by CFQ-11 | Baseline, Week 6, 12, 18 and 26

CONTACTS AND LOCATIONS:
Locations (1):
- Myrak Research Center, Miami Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
All information supplied by StemCyte, Inc in connection with this study and not previously published, is considered confidential information. This information includes, but is not limited to, the Investigator's Brochure, clinical protocol, case report forms and other scientific data. All data collected during the study are confidential. This confidential information shall remain the sole property of StemCyte, Inc, shall not be disclosed to others without the written consent of StemCyte, Inc, and shall not be used except in the performance of this study.

REFERENCES:
- [Derived] Huang YW, Chen YC, Lun Lau EY, Su YC, Tai LK, Rosenthal J, Wang J, Lee TY. REGENECYTE cord blood cell therapy in post-COVID syndrome: a phase IIa randomized, placebo-controlled trial. EClinicalMedicine. 2026 Jan 9;91:103737. doi: 10.1016/j.eclinm.2025.103737. eCollection 2026 Jan. PMID 41625963